CLINICAL TRIAL: NCT01414764
Title: Does Autologous Conditioned Plasma Enhance Rotator Cuff Tendon Healing After Surgery? A Radomized Control Trial.
Brief Title: Does Autologous Conditioned Plasma Enhance Rotator Cuff Tendon Healing After Surgery?
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The University of Western Australia (Other)
Collaborators: Arthrex, Inc. (Industry)
Responsible Party: Principal Investigator, Allan Wang, Clinical Professor of Orthopaedic Surgery, The University of Western Australia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11/75
Record Dates: First submitted 2011-06-23; First posted 2011-08-11 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Supraspinatus Tear
Keywords: rotator cuff tendon repair surgery; supraspinatus tendon repair

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Autologous conditioned plasma (ACP) (Active Comparator): 10ml of patient's own venous blood is aspirated. The syringe is centrifuged in a proprietary closed unit (Arthrex Medical Company) for 5 minutes. The red blood cells will be discarded, and the supernatant containing ACP (with additional CaCl to activate the ACP and local anaesthetic) is injected into the tendon bone junction and adjacent area under ultrasound guidance. No adverse consequences are anticipated by using the Arthrex ACP injection.
  * First injection at approximately 10 days post-operatively
  * Second Injection at approximately 21 days post-operatively
  Other Names:
  Platelet rich plasma (PRP)
  Interventions: Other: Autologous conditioned plasma (ACP)
- Placebo (Placebo Comparator): 10ml of patient's own venous blood is aspirated. The syringe is centrifuged in a proprietary closed unit (Arthrex Medical Company) for 5 minutes. The venous blood sample will be discarded and a placebo (saline + local anaesthetic) is injected to the surrounding tissue, but not into the tendon, under guided ultrasound.
  * First injection at approximately 10 days post-operatively
  * Second Injection at approximately 21 days post-operatively
  Interventions: Drug: Placebo

INTERVENTIONS:
Other: Autologous conditioned plasma (ACP) — 10ml of patient's own venous blood is aspirated. ACP (1ml) (extracted from centrifuged venous sample), with additional calcium chloride is then injected into the tendon-bone junction and adjacent area under guided ultrasound.
  * First injection at approximately 10 days post-operatively
  * Second Injection at approximately 21 days post-operatively
  Other Names: Platelet rich plasma (PRP)
  Arms: Autologous conditioned plasma (ACP)
Drug: Placebo — 10ml of patient's own venous blood is aspirated. The syringe is centrifuged in a proprietary closed unit (Arthrex Medical Company) for 5 minutes. The venous blood sample will be discarded and a placebo (1ml saline + local anaesthetic) is injected to the surrounding tissue, but not into the tendon, under guided ultrasound.
  * First injection at approximately 10 days post-operatively
  * Second Injection at approximately 21 days post-operatively
  Arms: Placebo

SUMMARY:
The aim of this study is to establish if the application of autologous conditioned plasma (ACP), also described as platelet rich plasma (PRP), to the site of supraspinatus tendon repair beginning within two weeks of surgery, can improve patient outcomes over the course of 12 months. These outcomes will be measured by post-surgical pain and function scores, shoulder strength and range of motion (ROM), and radiological parameters of tendon healing. Outcome measures will be compared to a control group of patients receiving placebo injections following surgery (saline plus local anaesthetic).

This study is significant for being the first double blind randomised control trial, using two PRP injections to examine the efficacy of a PRP preparation following surgical repair of supraspinatus tendon. The objective is to prolong and enhance the tendon healing response initiated by surgery.

The research hypothesis is that enhanced tendon healing following the PRP injections will lead to more rapid rehabilitation and lower rates of re-rupture of the repaired tendon compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50-75 years;
* In a non-dependent relationship;
* Full-thickness supraspinatus tendon tear (deemed repairable);
* Pre-operative platelet count greater than 150 000.

Exclusion Criteria:

* Previous rotator cuff repair surgery;
* Active/distal infection;
* Metabolic bone or blood disorders;
* Pre-existing conditions associated with upper extremity pain;
* Rotator cuff tears secondary to fracture;
* Prior ACP/PRP injections;
* Non-surgical rotator cuff treatment in the past month, including corticosteroids and anti-inflammatory treatment.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-05; Primary Completion 2015-01 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Changes in magnetic resonance imaging (MRI) score over time | Pre-operatively, and 12 months post-operatively
  MRI will assess the dimensions of the supraspinatus tear pre-operatively. MRI will assess the tendon healing of the supraspinatus tendon post-operatively at 12 months

SECONDARY OUTCOMES:
Changes in shoulder range of motion over time | pre-operatively, 3 months post-operatively, 6 months post-operatively, 12 months post-operatively
  Shoulder range of motion measures will include:
  * internal humeral rotation of the affected arm
  * external humeral rotation of the affected arm
  * forward flexion of the affected arm
  * abduction of the affected arm
Changes in strength of the shoulder musculature over time | 6 months post-operatively, 12 months post-operatively
  Muscular strength will be measured through:
  * internal humeral rotation of the affected arm
  * external humeral rotation of the affected arm
  * forward flexion of the affected arm
  * abduction of the affected arm
Changes in the visual analogue scale (VAS) for pain over time | Pre-operatively, 1st injection post-operatively, 2nd injection post-operatively, 6 weeks post-operatively, 12 weeks post-operatively, 6 months post-operatively, 12 months post-operatively
  The VAS is a scale from 1 to 10 and requires the patient to rate their pain along the scale; with 0 equating to no pain and 10 equating to the worst possible pain.
Changes in the Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) questionnaire over time | Pre-operatively, 6 weeks post-operatively, 12 weeks post-operatively, 6 months post-operatively, 12 months post-operatively
  The QuickDASH is a shortened version of the Disabilities of the Arm Shoulder and Hand (DASH) outcome measure. It uses 11 items instead of the original 30 items to measure physical function and symptoms in persons with any or multiple musculoskeletal disorders of the upper arm.
Changes in the Oxford Shoulder Score (OSS) over time | Pre-operatively, 6 weeks post-operatively, 12 weeks post-operatively, 6 months post-operatively, 12 months post-operatively
  The OSS is a self-reported questionnaire developed to evaluate disability in those with injuries and impairment of the rotator cuff.
Changes in the Simple Shoulder Test (SST) over time | Pre-operatively, 6 weeks post-operatively, 12 weeks post-operatively, 6 months post-operatively, 12 months post-operatively
  The SST consists of a series of 12 "yes" or "no" questions regarding function of the involved shoulder.
Changes in the Short Form - 12 health questionnaire (SF-12) over time | Pre-operatively, 6 weeks post-operatively, 12 weeks post-operatively, 6 months post-operatively, 12 months post-operatively
  The SF-12 is a shortened version of the Short Form-36 (SF-36). It uses 12 items instead of 36, to measure general functional health and well-being from the patient's point of view.

CONTACTS AND LOCATIONS:
Overall Officials: Allan Wang, FRACS PhD, Principal Investigator — The University of Western Australia; Timothy Ackland, BSc PhD, Study Chair — The University of Western Australia
Locations (1):
- Fremantle Hospital Radiology Department, Fremantle, Western Australia, Australia

REFERENCES:
- [Result] Randelli P, Arrigoni P, Ragone V, Aliprandi A, Cabitza P. Platelet rich plasma in arthroscopic rotator cuff repair: a prospective RCT study, 2-year follow-up. J Shoulder Elbow Surg. 2011 Jun;20(4):518-28. doi: 10.1016/j.jse.2011.02.008. PMID 21570659